CLINICAL TRIAL: NCT06613516
Title: CaptAin - Effect of Capivasertib on ctDNA in ER Positive Breast Cancer
Brief Title: Effect of Capivasertib on ctDNA in ER Positive Breast Cancer
Acronym: CaptAin
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was stopped because funder pulled funding for the study. 2 patients were screened however none of the screen patients were eventually recruited
Sponsor: Imperial College London (Other)
Collaborators: AstraZeneca (Industry); Sharp (Industry); Natera, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22CX7530; 2022-000802-82 (EudraCT Number)
Record Dates: First submitted 2024-08-19; First posted 2024-09-26 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer; Oestrogen Receptor Positive Breast Cancer
Keywords: Breast Cancer; Oestrogen receptor positive breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — capivasertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Subject to be dose with Capivasertib bidaily (Experimental): 400mg of Capivasertib to be dosed to patients and taken twice a day for a maximum of two years
  Interventions: Drug: Capivasertib

INTERVENTIONS:
Drug: Capivasertib — Capivasertib is a selective inhibitor of the kinase activity of the serine/threonine Akt/PKB pathway that may potentially provide clinical benefit over a range of therapeutic indications. Capivasertib comes in capsule form in two forms; 160mg or 200mg

SUMMARY:
There is growing evidence that cancer DNA (called circulating tumour DNA - ctDNA) in the blood is often an early sign that the cancer is likely to return. The aim of this study is to investigate whether treating women who have detectable ctDNA in their blood with a drug called Capivasertib can help control ctDNA levels and prevent developing metastatic or secondary breast cancer.

A recruitment of 20 women with oestrogen receptor (ER) positive breast cancer (who are already on standard of care hormone therapy who are being treated with curative intent) is aimed for; which means that the disease has not yet spread to distant parts of the body. Each subject will be dosed with 400mg of Capivasertib twice a day for a maximum period of two years.

DETAILED DESCRIPTION:
Early stage (I-III) ER positive HER2 negative breast cancer is treated with intensive multi-modal treatment which may include chemotherapy, radiotherapy and endocrine therapy given with curative intent. In spite of this, 10-40% of patients will ultimately relapse with incurable metastatic disease which will be terminal and life limiting. There is therefore a need to identify which patients are more at risk of relapse and develop strategies to alter the disease course in these patients.

There is a now a body of evidence that circulating tumour DNA (ctDNA) can be detected in the blood of patients who are going to relapse and that detection of this ctDNA antecedes clinical recurrence by approximately 9 months (Coombes et al, Garcia-Murillas et al).

This presents an ideal circumstance in which to intervene by considering ctDNA positive patients to have micrometastatic disease/molecular relapse and treating them with agents designed to modify the otherwise predictable outcome of relapse and ultimately death from their disease.

Capivasertib is a potent, selective inhibitor of the kinase activity of the serine/threonine Akt/PKB (protein kinase B) that is being developed as a potential treatment for solid and haematological malignancies. AZD5363 inhibits all three Akt isoforms and therefore has the potential to provide clinical benefit over a range of therapeutic indications.

Given the recent success of Capivasertib in extending progression free survival in metastatic ER positive breast cancer (FAKTION trial: Jones et al) it is proposed that treating ctDNA positive patients with this drug at this earlier stage may influence ctDNA levels and potentially the outcomes for these patients.

It is porposed to identify a cohort of ctDNA positive patients and treat them with Capivasertib and monitor their ctDNA levels prospectively over time whilst following the patients for toxicity and clinical outcomes.

Given that ctDNA positivity in ER positive breast cancer portends relapse whether Capivasertib affects ctDNA levels in patients who have detectable ctDNA will be established. Moreover, there is limited data on how ctDNA levels change over time especially in response to treatments and this study will offer valuable insights into that area which can feed into larger studies in the near future.

It is proposed to screen a number of patients who have completed standard of care curative intent treatment for their ER positive breast cancer and are established on aromatase inhibitor therapy (>6 months) and are planned to have ongoing endocrine therapy for at least another two years. Patients meeting the inclusion criteria will be screened until 20 ctDNA positive patients have been enrolled. The plan is to take blood at a single time point for each patient and will screen for ctDNA positivity using a personalised ctDNA assay as previously described (Coombes et al, Garcia-Murillas et al). Commercially available Signatera assay will be used to determine ctDNA positivity. Patients who are found to be ctDNA positive will then be started on treatment with Capivasertib and ctDNA levels will be followed over time. If patients are ctDNA negative on their first ctDNA sample they will have an opportunity to be re-tested for ctDNA every 3 months until the end of the screening period (which will end once 20 patients are recruited to start treatment). This is based on data that shows that ctDNA positivity pick-up rate improves with serial testing in patients over time (Coombes et al).

The hypothesis is that treating these ctDNA positive patients with Capivasertib will have an effect on the dynamics of the ctDNA measurements. Patients will also be followed over time to assess toxicity and acceptability of the drug and to monitor for overt metastatic relapse.

The outcome measures of the study is:

To monitor ctDNA dynamics during treatment with Capivasertib

* Percentage of patients with ctDNA clearance compared to baseline
* Duration of ctDNA clearance
* Percentage of patients with >50% decrease in ctDNA mean variant allele frequency (VAF) compared to baseline

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent prior to any study specific procedures
2. Female aged >18 years
3. Histologically confirmed ER positive HER2 negative breast cancer
4. Post menopausal (or biochemically post-menopausal)
5. Completed standard initial treatment and established on aromatase inhibitor (AI) for > 6 months and planned for at least 2 more years
6. Tolerating AI well
7. Eastern Cooperative Oncology Group (ECOG) performance status 0-1 (see Appendix 1) with no deterioration over the previous 2 weeks prior to baseline or day of first dosing
8. Minimum life expectancy of 12 weeks
9. Availability of tissue from diagnosis/treatment to assess ctDNA status
10. Relatively high risk for relapse (all except T1N0 or T2N0) using a risk stratified recruitment process
11. Adequate organ and bone marrow function as follows (a-c cannot be met with transfusions or growth factor support administered within 14 days of starting the first dose):

    1. Haemoglobin ≥9.0 g/dL (>5.59 mmol/L).
    2. Absolute neutrophil count ≥1.0×109/L.
    3. Platelet count ≥100×109/L.
    4. Total bilirubin ≤1.5×the upper limit of normal (ULN) or ≤3×ULN in the presence of documented Gilbert's syndrome (unconjugated hyperbilirubinemia).
    5. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≤2.5×ULN; for participants with hepatic metastases, ALT or AST ≤5×ULN.Elevated alkaline phosphatase (ALP) is not exclusionary if due to the presence of bone metastasis and liver function is otherwise considered adequate in the investigator's judgement.
    6. f) Creatinine clearance (CrCL) >50 mL/min per the Cockcroft-Gault formula (using actual body weight) without the need for chronic dialysis therapy.

Exclusion Criteria:

1. Metastatic disease at screening
2. ECOG performance status >1 (see Appendix 1)
3. History of another primary malignancy except for malignancy treated with curative intent with no known active disease ≥ 5 years before the first dose of study intervention and of low potential risk for recurrence. Exceptions include basal cell carcinoma of the skin and squamous cell carcinoma of the skin that has undergone potentially curative therapy
4. Known to have active hepatitis infection, positive hepatitis C antibody, hepatitis B virus surface antigen or hepatitis B virus core antibody, at screening. Known to have human immunodeficiency virus (HIV) with a CD4+ T-cell count < 350 cells/uL or a history of an acquired immunodeficiency syndrome (AIDS)-defining opportunistic infection within the past 12 months. (HIV inclusion criteria may be adjusted to lower CD4+ count values if clinically indicated if the patient has a potentially curable malignancy or for interventions in a later stage of development that have demonstrated prior activity within a given cancer, please adjust if necessary.) Known to have active tuberculosis infection (clinical evaluation that may include clinical history, physical examination and radiographic findings, or tuberculosis testing in line with local practice)
5. Known history of drug or alcohol abuse within 2 years
6. History of interstitial lung disease
7. Any other disease, physical examination finding, or clinical laboratory finding that, in the investigator's opinion, gives reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug, may affect the interpretation of the results, render the patient at high risk from treatment complications or interferes with obtaining informed consent
8. Clinically significant abnormalities of glucose metabolism as defined by any of the following at screening:

   1. Patients with diabetes mellitus type I or diabetes mellitus type II requiring insulin treatment
   2. HbA1c ≥ 8.0% (63.9 mmol/mol)
9. Prior treatment with any of the following:

   1. Participation in another clinical study with an IMP administered in the last <<2 weeks or 5 half-lives, whichever is longer
   2. AKT, PI3K and MTOR inhibitors
   3. Any other chemotherapy, immunotherapy, immunosuppressant medication (other than corticosteroids) or anticancer agents (other than current endocrine therapy with AI +/- LHRH analogies) within 3 weeks of the first dose of study treatment. A longer washout may be required for drugs with a long half-life (eg biologics) as agreed with the sponsor
   4. Palliative radiotherapy within 2 weeks; or radiotherapy to more than 30% of the bone marrow within 4 weeks before the first dose of study intervention
   5. Major surgical procedure (excluding placement of vascular access) or significant traumatic injury within 4 weeks of the first dose of study intervention or an anticipated need for major surgery during the study
   6. Potent inhibitors or inducers of CYP3A4 within 2 weeks prior to the first dose of study treatment (3 weeks for St John's Wort) or sensitive substrates of CYP344, CYP2C9 and/or CYP2D6 with a narrow therapeutic window within 1 week prior to the first study dose
10. Currently pregnant or breast feeding
11. As judged by the investigator, any evidence of diseases (such as severe or uncontrolled systemic diseases, including uncontrolled hypertension, renal transplant and active bleeding diseases which, in the investigator's opinion, makes it undesirable for the participant to participate in the study or that would jeopardise compliance with the protocol
12. Judgment by the investigator that the participant should not participate in the study if the participant is unlikely to comply with study procedures, restrictions and requirements
13. Participants with a known hypersensitivity to Capivasertib or any of the excipients of the product
14. Refractory nausea and vomiting, chronic gastrointestinal disease, inability to swallow the formulated product, or previous significant bowel resection that would preclude adequate absorption, distribution, metabolism, or excretion of Capivasertib
15. Persistent toxicities (CTCAE Grade ≥2) caused by previous anticancer therapy, excluding alopecia. Participants with irreversible toxicity that is not reasonably expected to be exacerbated by study intervention may be included (e.g. hearing loss)
16. Investigator judgment of 1 or more of the following:
17. Mean resting corrected QT interval >470 ms, obtained from ECG performed at screening.
18. Medical history significant for arrhythmia (e.g., multifocal premature ventricular contractions, bigeminy, trigeminy, ventricular tachycardia), which is symptomatic or requires treatment (CTCAE Grade 3), symptomatic or uncontrolled atrial fibrillation despite treatment, or asymptomatic sustained ventricular tachycardia. Participants with atrial fibrillation controlled by medication or arrhythmias controlled by pacemakers may be permitted to enter the study.
19. Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalaemia of Grade ≥1, potential for Torsades de Pointes, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age in first-degree relative, history of QT prolongation associated with other medications that required discontinuation of the medication (see section 6.5 for guidance on participants receiving any concomitant medication known to prolong the QT interval).
20. Experience of any of the following procedures or conditions in the preceding 6 months: coronary artery bypass graft, angioplasty, vascular stent, myocardial infarction, angina pectoris, congestive heart failure New York Heart Association (NYHA) grade ≥2.
21. Uncontrolled hypotension: systolic blood pressure <90 mmHg and/or diastolic blood pressure <50 mmHg.
22. Involvement in the planning and/or conduct of the study (applies to both Investigator staff and/or staff at the study site)
23. Previous enrolment in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Study is limited to biological females as this study is investigating breast cancer therapeutics
Enrollment: 0 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-09-16 (Actual); Study Completion 2025-09-16 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with complete ctDNA clearance | 2 years
  To monitor ctDNA dynamics during treatment with Capivasertib based on the percentage of patients with ctDNA clearance compared to baseline
Duration of ctDNA clearance | 2 years
  To monitor ctDNA dynamics during treatment with Capivasertib based on measuring the duration of ctDNA clearance
50% ctDNA clearance | 2 years
  To monitor ctDNA dynamics during treatment with Capivasertib based on the percentage of patients with over 50% decrease in ctDNA levels compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Dr Farah Rehman, Study Chair — Imperial College Healthcare Trust
Locations (1):
- Imperial College Healthcare Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Garcia-Murillas I, Schiavon G, Weigelt B, Ng C, Hrebien S, Cutts RJ, Cheang M, Osin P, Nerurkar A, Kozarewa I, Garrido JA, Dowsett M, Reis-Filho JS, Smith IE, Turner NC. Mutation tracking in circulating tumor DNA predicts relapse in early breast cancer. Sci Transl Med. 2015 Aug 26;7(302):302ra133. doi: 10.1126/scitranslmed.aab0021. PMID 26311728
- [Background] Jones RH, Casbard A, Carucci M, Cox C, Butler R, Alchami F, Madden TA, Bale C, Bezecny P, Joffe J, Moon S, Twelves C, Venkitaraman R, Waters S, Foxley A, Howell SJ. Fulvestrant plus capivasertib versus placebo after relapse or progression on an aromatase inhibitor in metastatic, oestrogen receptor-positive breast cancer (FAKTION): a multicentre, randomised, controlled, phase 2 trial. Lancet Oncol. 2020 Mar;21(3):345-357. doi: 10.1016/S1470-2045(19)30817-4. Epub 2020 Feb 5. PMID 32035020
- [Background] Coombes RC, Page K, Salari R, Hastings RK, Armstrong A, Ahmed S, Ali S, Cleator S, Kenny L, Stebbing J, Rutherford M, Sethi H, Boydell A, Swenerton R, Fernandez-Garcia D, Gleason KLT, Goddard K, Guttery DS, Assaf ZJ, Wu HT, Natarajan P, Moore DA, Primrose L, Dashner S, Tin AS, Balcioglu M, Srinivasan R, Shchegrova SV, Olson A, Hafez D, Billings P, Aleshin A, Rehman F, Toghill BJ, Hills A, Louie MC, Lin CJ, Zimmermann BG, Shaw JA. Personalized Detection of Circulating Tumor DNA Antedates Breast Cancer Metastatic Recurrence. Clin Cancer Res. 2019 Jul 15;25(14):4255-4263. doi: 10.1158/1078-0432.CCR-18-3663. Epub 2019 Apr 16. PMID 30992300
- [Background] Pan H, Gray R, Braybrooke J, Davies C, Taylor C, McGale P, Peto R, Pritchard KI, Bergh J, Dowsett M, Hayes DF; EBCTCG. 20-Year Risks of Breast-Cancer Recurrence after Stopping Endocrine Therapy at 5 Years. N Engl J Med. 2017 Nov 9;377(19):1836-1846. doi: 10.1056/NEJMoa1701830. PMID 29117498